CLINICAL TRIAL: NCT06071039
Title: Development of a 3D Spacer Mattress for Pressure Relieving in Cardiac Surgery and Evaluation of Its Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: İsmail TOYGAR (Other)
Collaborators: Bahçeşehir University (Other)
Responsible Party: Sponsor-Investigator, İsmail TOYGAR, Associate Professor, Ege University
Organization: Ege University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Bahcesehir
Record Dates: First submitted 2023-09-23; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Pressure Ulcer; Cardiac Surgery
Keywords: Pressure ulcer; Operating room; Cardiac Surgery
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: There were two groups in the trial. The first group was the group in which the patients used the mattress developed by the researcher. This was the intervention group. In the second group, the patients used the standard operating theatre mattress. This was the control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D Spacer Mattress (Experimental): For the patients in this group, the mattress which developed by the researchers was used. Pressure level between the body and the mattress was measured throughout the surgery.
  Interventions: Combination Product: 3D spacer Fabric Based Mattress
- Operating Room Mattress (No Intervention): For the patients in this group, the mattress which was in common use was used. The mattress used for the patients in this group was made up of foam. The pressure level between the body and the mattress was measured throughout the surgery.

INTERVENTIONS:
Combination Product: 3D spacer Fabric Based Mattress — For the patients in the intervention group, the 3D spacer fabric-based mattress was used instead of the operating room theater mattress. The pressure level of the patients was monitored throughout the surgery.
  Arms: 3D Spacer Mattress

SUMMARY:
In this study, researchers developed a mattress made of 3D spacer fabric to relieve pressure during cardiovascular surgery. Following the development process, an initial assessment of the mattress's effectiveness was carried out on healthy volunteers. The same people lay first on the developed product and then on the surgical mattress in the supine position. In both cases, the pressure between the person and the mattress was measured using a force-sensitive resistor (using Interlink's FRS-406 series sensors). Thirty patients were included in the initial evaluation. A randomised controlled trial was then carried out with patients undergoing surgery (patients were divided into two groups; (a) mattress developed by the researchers and (b) standard operating theatre mattress). Sixty patients were divided into two groups using block randomisation. In the block randomisation, patients below or above body mass index 27 were equally distributed between the groups. Pressure levels were measured continuously during surgery using the same sensors.

DETAILED DESCRIPTION:
In this study, the researchers developed a mattress made of 3D spacer fabric for pressure relief during cardiovascular surgery. Following the development process, an initial assessment of the mattress's effectiveness was carried out on healthy volunteers. The same people lay first on the developed product and then on the surgical mattress in the supine position. In both cases, the pressure between the person and the mattress was measured using a force-sensitive resistor (using Interlink's FRS-406 series sensors). 30 patients were included in the initial evaluation. A randomised controlled trial was then carried out with patients who underwent surgery (patients were divided into two groups; (a) mattress developed by the researchers and (b) operating theatre mattress in common use). 60 patients were divided into two groups using block randomisation. In the block randomisation, patients below or above body mass index 27 were evenly distributed between the groups. Pressure levels were continuously measured during surgery using the same sensors. Data were analysed using IBM SPSS software v26.

ELIGIBILITY:
Inclusion criteria:

* Being 18 years or older
* Not having a pressure ulcer prior to surgery
* Agreeing to participate in the study

Exclusion criteria:

- Not agreeing to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Pressure level | through study completion, an average of 1 yea
  Pressure between the product surface and patients' body

CONTACTS AND LOCATIONS:
Overall Officials: ismail toyğar, Ph.D., Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Şehit Prof. Dr. İlhan Varank Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Isler Isildak Y, Eti Aslan F, Korkmaz E, Comez L, Toygar I. Development of a Three-dimensional Spacer Mattress for Pressure Relief in Cardiac Surgery and Evaluation of Its Efficacy: A Feasibility Study. Adv Skin Wound Care. 2025 Nov-Dec 01;38(10):547-555. doi: 10.1097/ASW.0000000000000368. Epub 2025 Sep 30. PMID 41037744